CLINICAL TRIAL: NCT05703334
Title: Kinesio Tape Versus Myofascial Release of Respiratory Muscles on Athletes Performance With Exercise Induced Asthma
Brief Title: Kt and Myofascial Release in Exc Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled mohammed Ahmed zaki, Dr khaled zaki, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/003279
Record Dates: First submitted 2023-01-16; First posted 2023-01-30 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Exercise Induced Asthma
Keywords: Pulmonary function test
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: seventy male athletic subjects with exercise induced asthma, their age ranged from 18-30 years old in this study , with group (A) mean age (21.03+3.6 years), and mean BMI values (27.6+.9 kg/m2) ,and group (B) mean age (21.9+3.8 years),and mean BMI values (27.8+1.3 kg/m2), and group (C) mean age(22+3.1 years), and mean BMI values (27.8+1.3 kg/m2).
  Subjects were assigned randomly into tow study groups and one control group:Group(A) 30 subjects were treated by kinesio tap therapy 2sessions per week,Ground(B) 30 subjects were treated by myofascial release therapy 3 sessions per week ,Group (C) 10 subjects were not recieved treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio tap (Experimental): group (A) mean age (21.03+3.6 years), and mean BMI values (27.6+.9 kg/m2 Group(A) 30 subjects were treated by kinesio tap therapy 2sessions per week.
  Interventions: Other: Kinesio tap
- Myofascial release (Experimental): group (B) mean age (21.9+3.8 years),and mean BMI values (27.8+1.3 kg/m2 Ground(B) 30 subjects were treated by myofascial release therapy 3 sessions per week .
  Interventions: Other: Kinesio tap
- Control group (No Intervention)

INTERVENTIONS:
Other: Kinesio tap — Applied on pulmonary muscles :diaphragm muscle and abdominal muscle and sternocleinomastoid muscle 3 time per weak for 2 mounth
  Other Names: Myofascial release
  Arms: Kinesio tap; Myofascial release

SUMMARY:
Purpose of this study was to compare between the effects of kinesio tap and myofascial release of respiratory muscles on exercise induced asthma

DETAILED DESCRIPTION:
seventy male athletic subjects with exercise induced asthma, their age ranged from 18-30 years old in this study , with group (A) mean age (21.03+3.6 years), and mean BMI values (27.6+.9 kg/m2) ,and group (B) mean age (21.9+3.8 years),and mean BMI values (27.8+1.3 kg/m2), and group (C) mean age(22+3.1 years), and mean BMI values (27.8+1.3 kg/m2).

Subjects were assigned randomly into tow study groups and one control group:Group(A) 30 subjects were treated by kinesio tap therapy 2sessions per week,Ground(B) 30 subjects were treated by myofascial release therapy 3 sessions per week ,Group (C) 10 subjects were not recieved treatment.

ELIGIBILITY:
Inclusion Criteria:

* Seventy male athlete with ages ranging from 18 to 28 years old. Their Body Mass Index ranged from "18.5" to "24.9". They have the same level of good aerobic fitness, muscular strength and endurance, and flexibility according to tests results; running or jogging test, push up or sit up test, and sit-and-reach test respectively.

Exclusion Criteria:

1. Pulmonary disorders.
2. Metabolic disorders (e.g. Diabetes Mellitus).
3. Coronary artery disorders .
4. Neurological disorders.
5. Recent musculoskeletal injuries.
6. Renal disorders.
7. Hepatic disorders.
8. Skin hypersensitive.
9. Smokers

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test | 2 months
  MVV :liter FVC:liter FEV1:liter FVC/FEV1:% VC:liter

SECONDARY OUTCOMES:
Cooper's 12 minute run test | 2 months
  Vo2 max:ml/kg/min

OTHER OUTCOMES:
pulse oximeter | 2 months
  Pao2:%
IFIS | 2 months
  General fitness

CONTACTS AND LOCATIONS:
Locations (1):
- Khaled mohamed Ahmed zaki, Port Said, Port Said/el Manakh, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://doi.org/10.1038/s41533-018-0098-2
- See also: Related Info — http://doi.org/10.1183/20734735.008116